CLINICAL TRIAL: NCT04388254
Title: A 12-Month, Open-Label Safety Study of Simufilam Followed by a 6-Month Randomized Withdrawal and 6 Additional Months Open-Label in Mild-to-moderate Alzheimer's Disease Patients
Brief Title: Simufilam (PTI-125), 100 mg, for Mild-to-moderate Alzheimer's Disease Patients
Acronym: PTI-125
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cassava Sciences, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-125-04; R44AG065152 (NIH)
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam; Tablets

STUDY DESIGN:
Intervention Model Description: Approximately two hundred (200) patients will be enrolled into the study. All participants will receive open-label simufilam 100 mg b.i.d. for a year. At Month12, participants will be randomized (1:1) to continue taking simufilam 100 mg b.i.d. or to be switched to placebo for 6 months. At Month 18, all participants will enter a final 6-month treatment period of open-label simufilam 100 mg b.i.d.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo for the 6-month randomized period (Month 12 to Month 18)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Simufilam 100 mg oral tablets throughout (Experimental): Simufilam 100 mg oral tablets administered twice daily (BID) for the full 24 months (including the randomized period Month 12 to Month 18)
  Interventions: Drug: Simufilam 100 mg oral tablet
- Simufilam 100 mg oral tablets / Placebo / Simufilam 100 mg oral tablets (Placebo Comparator): This placebo arm is only for Month 12 to Month 18. Day 1 to Month 12, as well as Month 18 to Month 24 are open-label treatment periods of simufilam 100 mg b.i.d. for all subjects.
  Interventions: Drug: Simufilam 100 mg oral tablet; Drug: Placebo

INTERVENTIONS:
Drug: Simufilam 100 mg oral tablet — Simufilam 100 mg oral tablet for b.i.d. administration
  Other Names: PTI-125; Sumifilam
Drug: Placebo — Matching placebo oral tablets
  Arms: Simufilam 100 mg oral tablets / Placebo / Simufilam 100 mg oral tablets

SUMMARY:
A two-year safety study of simufilam (PTI-125) 100 mg oral tablets twice daily for participants of the previous simufilam studies as wells as additional new mild-to-moderate Alzheimer's disease subjects for a total of 200 participants. All participants will receive simufilam 100 mg tablets twice daily for one year, followed by a 6-month randomized, double-blind period where subjects will either continue on active treatment or be switched to placebo. The study concludes with an additional 6-month open-label treatment period. Clinic visits are every month or month and a half in the first year, and every 3 months in the second year with an additional visit at Month 13. Cognition and neuropsychiatric symptoms are evaluated.

DETAILED DESCRIPTION:
The objectives of this study are to build the safety database for simufilam (PTI-125) and to investigate its effects on biomarkers, cognition and neuropsychiatric symptoms during 12-month twice-daily administration in mild-to-moderate AD patients. Additional objectives are to assess differences in cognition and neuropsychiatric symptoms between active and placebo arms in the 6-month randomized period. All subjects will undergo lumbar puncture at screening for baseline testing of cerebrospinal fluid (CSF) total tau and Abeta42, and the first 50 subjects will also provide a CSF sample at Month 6 or Month 12 for evaluation of change from baseline in CSF biomarkers. CSF will not be required of subjects with prior CSF, PET or MRI evidence of Alzheimer's disease. Plasma biomarkers will be evaluated in all subjects. Safety will be assessed by blood tests, electrocardiograms, adverse event monitoring and, at Months 12 and 24, full physical examinations.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Informed consent form (ICF) signed by the subject or legally acceptable representative.
2. Patient has a caregiver or legal representative responsible for administering the drug and recording the time.
3. Ages ≥ 50 and ≤ 85 years
4. Clinical diagnosis of dementia due to possible or probable AD consistent with criteria established by a workgroup of the National Institute on Aging and the Alzheimer's Disease Association.
5. If female, postmenopausal for at least 1 year
6. Patient living at home, senior residential setting, or an institutional setting without the need for continuous (i.e. 24-h) nursing care
7. General health status acceptable for participation in the study
8. Fluency (oral and written) in English or Spanish
9. If receiving memantine, rivastigmine, galantamine or an AChEI, receiving a stable dose for at least 3 months (90 days) before screening. If receiving donepezil, receiving any dose lower than 23 mg once daily. Multiple medications are allowed.
10. The patient is a non-smoker for at least 3 years.
11. The patient or legal representative must agree to comply with the drawing of blood samples for the PK assessments, laboratory assessments and SavaDx.
12. MMSE-2 score ≥ 16 and ≤ 26 at screening, OR if > 26, must have evidence of AD pathology such as a prior CSF total tau/Aβ42 ratio ≥ 0.28, an amyloid positive PET scan or hippocampal volume loss consistent with AD.

EXCLUSION CRITERIA:

1. Anything that in the opinion of the Investigator would preclude participation in a 2-year study.
2. BMI < 18.5
3. Positive urine drug screen.
4. Positive HIV, HCV or HbsAg screen.
5. Suicidality on C-SSRS
6. Exposure to an experimental drug other than simufilam, experimental biologic or experimental medical device within 3 months before screening
7. A medical condition that would interfere with a lumbar puncture
8. Residence in a skilled nursing facility and requiring 24 h care.
9. Clinically significant laboratory test results
10. Clinically significant untreated hypothyroidism (if treated, thyroid-stimulating hormone level and thyroid supplementation dose must be stable for at least 6 months before screening)
11. Insufficiently controlled diabetes mellitus, including requiring insulin or metformin >1000 mg/day.
12. Renal insufficiency (serum creatinine > ULN and clinically significant in the opinion of PI and/or Sponsor OR eGFR <60 ml/min/m2 as estimated by either the MDRD or CKD-EPI equation)
13. Malignant tumor within 3 years before screening (except squamous and basal cell carcinoma or cervical carcinoma in situ or localized prostate cancer or localized stage 1 bladder cancer)
14. History of ischemic colitis or ischemic enterocolitis
15. Unstable medical condition that is clinically significant in the judgment of the investigator
16. Alanine transaminase (ALT) or aspartate transaminase (AST) > ULN or total bilirubin > ULN and clinically significant in the opinion of PI and/or Sponsor.
17. History of myocardial infarction or unstable angina within 6 months before screening
18. History of more than 1 myocardial infarction within 5 years before screening
19. Clinically significant cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (patients with a pacemaker are acceptable)
20. Symptomatic hypotension, or uncontrolled hypertension
21. Clinically significant abnormality on screening electrocardiogram (ECG), including but not necessarily limited to a confirmed QTc (Fridericia correction method) value ≥ 450 msec for males or ≥ 470 msec for females.
22. Stroke within 18 months before screening, or history of a stroke concomitant with onset of dementia
23. History of brain tumor or other clinically significant space-occupying lesion on CT or MRI
24. Head trauma with clinically significant loss of consciousness within 12 months before screening or concurrent with the onset of dementia
25. Onset of dementia secondary to cardiac arrest, surgery with general anesthesia, or resuscitation
26. Specific degenerative CNS disease diagnosis other than AD (e.g., Huntington's disease, Creutzfeld-Jacob disease, Down's syndrome, Frontotemporal Dementia, Parkinson's disease)
27. Wernicke's encephalopathy
28. Active acute or chronic CNS infection
29. Donepezil 23 mg or greater QD currently or within 3 months prior to randomization
30. Discontinued AChEI < 30 days prior to randomization
31. Antipsychotics; low doses are allowed only if given for sleep disturbances, agitation and/or aggression, and only if the subject has received a stable dose for at least 3 months before randomization
32. Tricyclic antidepressants and monoamine oxidase inhibitors; all other antidepressants are allowed only if the subject has received a stable dose for at least 3 months before randomization
33. Anxiolytics or sedative-hypnotics, including barbiturates (unless given in low doses for benign tremor); low doses of benzodiazepines and zolpidem are allowed only if given for insomnia/sleep disturbance, and only if the subject has received a stable dose for at least 3 months before randomization
34. Immunosuppressants, including systemic corticosteroids, if taken in clinically immunosuppressive doses (Steroid use for allergy or other inflammation is permitted.)
35. Antiepileptic medications if taken for control of seizures
36. Chronic intake of opioid-containing analgesics
37. Sedating H1 antihistamines
38. Nicotine therapy (all dosage forms including a patch), varenicline (Chantix), or similar therapeutic agent within 30 days before screening
39. Clinically significant illness within 30 days of enrollment
40. History of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease
41. Loss of a significant volume of blood (> 450 mL) within 4 weeks prior to the study
42. COVID-19 infection within 3 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burns, PhD, Study Chair — Cassava Sciences
Locations (17):
- United States (15):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - Cognitive Clinical Trials, Surprise, Arizona
  - Sun Valley Research Center, Inc., Imperial, California
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Optimus U, Miami, Florida
  - Adaptive Clinical Research, Inc, Miami Lakes, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Cognitive Clinical Trials, Bellevue, Nebraska
  - Cognitive Clinical Trials, Omaha, Nebraska
  - Advanced Memory Research Institute, Toms River, New Jersey
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Senior Adults Specialty Research, Austin, Texas
  - Centex Studies, Inc., Houston, Texas
  - Centex Studies, McAllen, Texas
- Canada (2):
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang HY, Pei Z, Lee KC, Lopez-Brignoni E, Nikolov B, Crowley CA, Marsman MR, Barbier R, Friedmann N, Burns LH. PTI-125 Reduces Biomarkers of Alzheimer's Disease in Patients. J Prev Alzheimers Dis. 2020;7(4):256-264. doi: 10.14283/jpad.2020.6. PMID 32920628
- [Background] Wang HY, Lee KC, Pei Z, Khan A, Bakshi K, Burns LH. PTI-125 binds and reverses an altered conformation of filamin A to reduce Alzheimer's disease pathogenesis. Neurobiol Aging. 2017 Jul;55:99-114. doi: 10.1016/j.neurobiolaging.2017.03.016. Epub 2017 Mar 31. PMID 28438486
- [Background] Wang HY, Bakshi K, Frankfurt M, Stucky A, Goberdhan M, Shah SM, Burns LH. Reducing amyloid-related Alzheimer's disease pathogenesis by a small molecule targeting filamin A. J Neurosci. 2012 Jul 18;32(29):9773-84. doi: 10.1523/JNEUROSCI.0354-12.2012. PMID 22815492
- [Derived] Brodtmann A, Darby D, Oboudiyat C, Mahoney CJ, Le Heron C, Panegyres PK, Brew B. Assessing preparedness for Alzheimer disease-modifying therapies in Australasian health care systems. Med J Aust. 2023 Apr 3;218(6):247-249. doi: 10.5694/mja2.51880. Epub 2023 Mar 19. No abstract available. PMID 36934371

RESULTS

PARTICIPANT FLOW:
Groups:
- Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease: Simufilam 100 mg oral tablets administered twice daily (BID); Subjects with a Mini Mental State Examination (MMSE) score of >=21 are included in Mild group
- Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease: Subjects with a Mini Mental State Examination (MMSE) score of >=21 are included in Mild group;
  The placebo arm is only from Month 12 to Month 18. Day 1 to Month 12, as well as Month 18 to Month 24 are open-label treatment periods of simufilam 100 mg b.i.d.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration;
  Placebo: Matching placebo oral tablets
- Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease: Simufilam 100 mg oral tablets administered twice daily (BID); Subjects with a Mini Mental State Examination (MMSE) score of <=20 are included in Moderate group
- Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease: Subjects with a Mini Mental State Examination (MMSE) score of <=20 are included in Moderate group;
  The placebo arm is only from Month 12 to Month 18. Day 1 to Month 12, as well as Month 18 to Month 24 are open-label treatment periods of simufilam 100 mg b.i.d.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
  Placebo: Matching placebo oral tablets
Period: Open Label Period 1 (Mth 1 to Mth 12)
Arm/Group | Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease | Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease | Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease | Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease
Started (All subjects started and were administered simufilam for the first 12 months) | 134 | 0 | 85 | 0
Completed 12 Months and Chose Not to Continue | 15 | 0 | 5 | 0
Discontinued Before Completing 12 Months | 30 | 0 | 13 | 0
Completed 12 Months and Chose to Continue | 104 | 0 | 72 | 0
Completed | 104 | 0 | 72 | 0
Not Completed | 30 | 0 | 13 | 0
Period: Double Blind Treatment (Mth12 to Mth18)
Arm/Group | Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease | Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease | Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease | Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease
Started | 48 | 41 | 32 | 35
Discontinued During Double Blind Treatment Period | 5 | 7 | 6 | 6
Completed | 43 | 34 | 26 | 29
Not Completed | 5 | 7 | 6 | 6
Period: Open Label Period 3 (Mth 18 to Mth 24)
Arm/Group | Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease | Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Mild Alzheimer's Disease | Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease | Simufilam 100 mg Oral Tablets/Placebo/Simufilam 100 mg Oral Tablets w/ Moderate Alzheimer's Disease
Started | 43 | 34 | 26 | 29
Discontinued During Period 3 | 4 | 0 | 4 | 3
Completed | 39 | 34 | 22 | 26
Not Completed | 4 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: It wouldn't make sense to provide updated demographic baseline information at the start of each period when only the participants age and BMI would differ with time. If there was a direct correlation to BMI and study drug, it would be reflected in the AE section or the safety section. One moderate subject was enrolled but was administered simufilam prior to day1 baseline efficacy procedures. That is why all data sets account for one less moderate subject.
Groups:
- Moderate Alzheimer's Disease: Subjects with a Mini Mental State Examination (MMSE) score of <=20 are included in Moderate group
- Mild Alzheimer's Disease: Subjects with a Mini Mental State Examination (MMSE) score of >=21 are included in Mild group
- Total: Total of all reporting groups
Arm/Group | Moderate Alzheimer's Disease | Mild Alzheimer's Disease | Total
Number analyzed (Participants) | 85 | 134 | 219
Age, Categorical [Count of Participants; unit: Participants] — Population: One moderate subject had their baseline MMSE collected after day 1 dose administration.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 22 | 26 | 48
    >=65 years | 63 | 108 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One moderate subject had their baseline MMSE collected after day 1 dose administration.
  years | 70.5 (8.7) | 70.8 (7.93) | 70.7 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One moderate subject had their baseline MMSE collected after day 1 dose administration.
  Participants
    Female | 55 | 68 | 123
    Male | 30 | 66 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One moderate subject had their baseline MMSE collected after day 1 dose administration.
  Participants
    Hispanic or Latino | 9 | 39 | 48
    Not Hispanic or Latino | 76 | 95 | 171
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One moderate subject had their baseline MMSE collected after day 1 dose administration.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 6 | 0 | 6
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 2 | 4 | 6
    White | 76 | 129 | 205
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m2] — Population: One moderate subject had their baseline MMSE collected after day 1 dose administration.
  kg/m2 | 25.52 (4.046) | 28.44 (5.740) | 27.33 (5.333)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ADAS-Cog-11
Description: Alzheimer's Disease Assessment Scale-Cognitive Subscale 11-item: Change from baseline in cognition over the course of 24 months Possible range in score: 0-70; Subscales are summed; Higher values represent a more cognitively impaired participant Decrease in mean value represents improvement in cognition from one timepoint to the next.
Time Frame: Day 1 to Month 24
Population: Full Analysis set; Overall number of participants is the number for each arm that completed a ADAS-Cog-11 assessment at baseline and month 24.
Measure: Mean (Standard Error); unit: Change in scale units
Groups:
- Moderate Alzheimer's Disease, 24 Months of Simufilam: * Moderate subjects: Mini Mental State Examination (MMSE) score of <=20
  * Subjects were administered Simufilam over the course of the whole trial (from day 1 to month 24)
- Mild Alzheimer's Disease, 24 Months of Simufilam: * Mild Subjects with a Mini Mental State Examination (MMSE) score of >=21
  * Subjects were administered Simufilam over the course of the whole trial (from day 1 to month 24)
- Moderate Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 18: * Moderate subjects: Mini Mental State Examination (MMSE) score of <=20
  * Subjects that were administered Simufilam from day 1 to month 12 and month 18 to 24 with 6 month simufilam interruption (placebo administration from month 12 to month 18)
- Mild Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 18: * Mild Subjects with a Mini Mental State Examination (MMSE) score of >=21
  * Subjects that were administered Simufilam from day 1 to month 12 and month 18 to 24 with 6 month simufilam interruption (placebo administration from month 12 to month 18)
Arm/Group | Moderate Alzheimer's Disease, 24 Months of Simufilam | Mild Alzheimer's Disease, 24 Months of Simufilam | Moderate Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 18 | Mild Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 18
Number analyzed (Participants) | 20 | 39 | 24 | 33
Change in scale units | 11.05 (1.19) | 0.07 (1.15) | 14.26 (1.79) | 1.04 (1.65)

2. Primary Outcome: Change From Baseline in ADAS-Cog-11 (Month 12 to Month 24)
Description: Alzheimer's Disease Assessment Scale-Cognitive Subscale 11-item: Change from baseline in cognition Starting at month 12 through month 24; Possible range in score: 0-70; Higher values represent a more cognitively impaired participant; Decrease in mean value represents improvement in cognition from one timepoint to the next.
Time Frame: Month 12 to Month 24
Population: Full Analysis set; Overall number of participants is the number for each arm/group that completed a ADAS-Cog-11 assessment at month 12 and month 24.
Measure: Mean (Standard Error); unit: Change in scale units
Groups:
- Moderate Alzheimer's Disease, 12 Months of Simufilam: * Moderate subjects: Mini Mental State Examination (MMSE) score of <=20
  * Subjects stayed on b.i.d. simufilam administration from month 12 through month 24 after already completing 12 months of b.i.d. simufilam administration
- Mild Alzheimer's Disease, 12 Months of Simufilam: * Mild Subjects with a Mini Mental State Examination (MMSE) score of >=21
  * Subjects stayed on b.i.d. simufilam administration from month 12 through month 24 after already completing 12 months of b.i.d. simufilam administration
- Moderate Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 24: * Moderate subjects: Mini Mental State Examination (MMSE) score of <=20
  * Subjects started 6 months of b.i.d. placebo administration at month 12 through month 18 after already completing 12 months of b.i.d. simufilam administration. Then re-started b.i.d. simufilam administration at month 18 for an additional 6 months.
- Mild Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 24: * Mild Subjects with a Mini Mental State Examination (MMSE) score of >=21
  * Subjects started 6 months of b.i.d. placebo administration at month 12 through month 18 after already completing 12 months of b.i.d. simufilam administration. Then re-started b.i.d. simufilam administration at month 18 for an additional 6 months.
Arm/Group | Moderate Alzheimer's Disease, 12 Months of Simufilam | Mild Alzheimer's Disease, 12 Months of Simufilam | Moderate Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 24 | Mild Alzheimer's Disease, Interrupted Simufilam Placebo Administration From Month 12 to Month 24
Number analyzed (Participants) | 19 | 35 | 23 | 30
Change in scale units | 7.39 (1.447) | 1.93 (1.128) | 6.97 (1.404) | 2.45 (1.225)

3. Primary Outcome: Safety and Tolerability (Open Label Abnormal Vital Signs)
Description: The most frequently reported Treatment Emergent Adverse Events indicative of abnormal vital signs (hypertension/worsening of hypertension and blood pressure increase) of simufilam (PTI-125) during the open label portion of the study: Open-label period 1 (Day 1 to Month 12) and open-label period 2 (Month 18 to Month 24)
Time Frame: Day 1 to Month 12 and month 18 to month 24
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Number of subjects that reported TEAEs while on Simufilam 100 mg oral tablets administered twice daily (BID) from Day 1 to month 12 and again from month 18 to month 24.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 171
Participants
  Hypertension/worsening hypertension | 13
  Blood pressure increase | 6
  The number of subjects that did not report hypertension or did not have worsening of hypertension | 152

4. Primary Outcome: Safety and Tolerability (Randomize Withdraw Abnormal Vital Signs)
Description: The most frequently reported Treatment Emergent Adverse Event indicative of abnormal vital signs (hypotension) of simufilam (PTI-125) or placebo during the randomized withdraw portion of the study : Month 12 to Month 18
Time Frame: Month 12 to month 18
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Number of subjects that reported TEAE indicative of abnormal vital signs (hypotension) while on Simufilam 100 mg oral tablets administered twice daily (BID) from month 12 to month 18.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
- Placebo: Number of subjects that reported TEAE indicative of abnormal vital signs (hypotension) while on placebo oral tablets administered twice daily (BID) from month 12 to month 18.
Arm/Group | Simufilam 100 mg Oral Tablets | Placebo
Number analyzed (Participants) | 45 | 37
Participants
  Number of subjects that reported hypotension | 2 | 0
  Number of subjects that did not report hypotension | 43 | 37

5. Primary Outcome: Safety and Tolerability (Open Label Electrocardiogram Results)
Description: The number of subjects that had Treatment Emergent Adverse Events indicative of abnormal Electrocardiogram results while on simufilam (PTI-125) during the open label portion of the study: Open-label period 1 (Day 1 to Month 12) and open-label period 2 (Month 18 to Month 24)
Time Frame: Day 1 to Month 12 and month 18 to month 24
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Number of subjects that reported TEAEs indicative of abnormal Electrocardiogram results while on Simufilam 100 mg oral tablets administered twice daily (BID) from Day 1 to month 12 and again from month 18 to month 24.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 171
Participants
  Acute left ventricular failure | 1
  Acute myocardial infarction | 3
  Angina pectoris | 2
  Aortic valve incompetence | 1
  Atrial fibrillation | 4
  Atrial tachycardia | 1
  Bradycardia | 3
  Cardiogenic shock | 1
  Coronary artery disease | 2
  Mitral valve incompetence | 2
  Sinus tachycardia | 1
  Subjects that reported TEAEs that were not related to Electrocardiogram results | 150

6. Primary Outcome: Safety and Tolerability (Randomize Withdraw Electrocardiogram Results)
Description: The number of subjects that had Treatment Emergent Adverse Events indicative of abnormal Electrocardiogram results while on simufilam (PTI-125) or placebo during the randomized withdraw portion of the study: Month 12 to Month 18
Time Frame: Month 12 to Month 18
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Number of subjects that reported TEAEs indicative of abnormal Electrocardiogram results while on Simufilam 100 mg oral tablets administered twice daily (BID) from month 12 to month 18.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
- Placebo: Number of subjects that reported TEAEs indicative of abnormal Electrocardiogram results while on placebo oral tablets administered twice daily (BID) from month 12 to month 18.
Arm/Group | Simufilam 100 mg Oral Tablets | Placebo
Number analyzed (Participants) | 45 | 37
Participants
  Acute Myocardial Infarction | 1 | 0
  Arrhymia | 0 | 1
  Atrial Fibrillation | 1 | 1
  Atrioventricular block first degree | 0 | 1
  Cardiomegaly | 0 | 1
  Subjects that had TEAEs that were not related Electrocadiogram results | 43 | 33

7. Primary Outcome: Safety and Tolerability (Open Label Abnormal Physical Examination)
Description: The most frequently reported Treatment Emergent Adverse Events indicative of abnormal physical examination (weight increase or weight decrease) while administered simufilam (PTI-125) during the open label portion of the study: Open-label period 1 (Day 1 to Month 12) and open-label period 2 (Month 18 to Month 24)
Time Frame: Day 1 to Month 12 and month 18 to month 24
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Number of subjects that reported TEAEs indicative of abnormal physical examination while on simufilam 100 mg oral tablets administered twice daily (BID) from Day 1 to month 12 and again from month 18 to month 24.
  Simufilam 100 mg oral tablet: simufilam 100 mg oral tablet for b.i.d. administration
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 171
Participants
  Weight decrease | 4
  Weight increase | 2
  Number of subjects that reported TEAEs not indicative of weight change | 165

8. Primary Outcome: Safety and Tolerability (Randomize Withdraw Abnormal Physical Examination Findings)
Description: The number of subjects that had Treatment Emergent Adverse Events of indicative of abnormal physical examination while on simufilam (PTI-125) or placebo during the randomized withdraw portion of the study: Month 12 to Month 18
Time Frame: Month 12 to Month 18
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Number of subjects that reported TEAEs indicative of abnormal physical examination while on Simufilam 100 mg oral tablets administered twice daily (BID) from month 12 to month 18.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
- Placebo: Number of subjects that reported TEAEs indicative of abnormal physical examination while on placebo oral tablets administered twice daily (BID) from month 12 to month 18.
Arm/Group | Simufilam 100 mg Oral Tablets | Placebo
Number analyzed (Participants) | 45 | 37
Participants
  Weight decrease | 0 | 2
  Subjects that did not report TEAEs of abnormal weight decrease | 45 | 35

9. Primary Outcome: Safety and Tolerability (Open Label Abnormal Clinical Laboratory Results)
Description: Treatment Emergent Adverse Events when three or more subjects reported abnormal clinical laboratory results while on simufilam (PTI-125) during the open label portion of the study: Open-label period 1 (Day 1 to Month 12) and open-label period 2 (Month 18 to Month 24)
Time Frame: Day 1 to Month 12 and month 18 to month 24
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: TEAEs when three or more subjects reported abnormal clinical laboratory results while on Simufilam 100 mg oral tablets administered twice daily (BID) from Day 1 to month 12 and again from month 18 to month 24.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 171
Participants
  Hyperkalaemia | 3
  Hyperlipidaemia | 3
  Hypophosphataemia | 3
  Subjects that reported 2 or less TEAEs indicative of clinical laboratory results | 162

10. Primary Outcome: Safety and Tolerability (Randomize Withdraw Abnormal Clinical Laboratory Results)
Description: Treatment Emergent Adverse Events when two or more subjects reported abnormal clinical laboratory results while on simufilam (PTI-125) or placebo during the randomized withdraw portion of the study: Month 12 to Month 18
Time Frame: Month 12 to Month 18
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg Oral Tablets: Treatment Emergent Adverse Events when two or more subjects reported abnormal clinical laboratory results while on Simufilam 100 mg oral tablets administered twice daily (BID) from month 12 to month 18.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
- Placebo: Treatment Emergent Adverse Events when two or more subjects reported abnormal clinical laboratory results while on placebo oral tablets administered twice daily (BID) from month 12 to month 18.
Arm/Group | Simufilam 100 mg Oral Tablets | Placebo
Number analyzed (Participants) | 45 | 37
Participants
  Leukocytosis | 0 | 2
  Haematuria | 2 | 1
  Two subjects or less that report TEAEs of abnormal clinical laboratory results or none at all. | 43 | 34

11. Secondary Outcome: Change From Baseline to Month 12 in Cerebral Spinal Fluid for Triggering Receptor Expressed on Myeloid Cells 2 (TREM2) Mean Concentration (pg/mL)
Description: Change from baseline to month 12 in Cerebral Spinal Fluid for Triggering Receptor Expressed on Myeloid Cells 2 (TREM2) Mean Concentration (pg/mL) (samples stored at -70 degrees Celsius; assays performed at Abilene Christian University Bioanalytics Laboratory)
Time Frame: Day 1 to Month 12
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Simufilam 100 mg Oral Tablets: Subjects administered Simufilam 100 mg oral tablets administered twice daily (BID) from Day 1 to month 12
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 13
pg/mL | -4093.31 (4730.736)

12. Secondary Outcome: Change From Baseline to Month 12 in Cerebral Spinal Fluid for Tau Protein Mean Concentration (pg/mL)
Description: Change from baseline to month 12 in Cerebral Spinal Fluid for Tau Protein Mean Concentration (pg/mL) (samples stored at -70 degrees Celsius; assays performed at Abilene Christian University Bioanalytics Laboratory)
Time Frame: Day 1 to Month 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 18
pg/mL | -12.26 (96.238)

13. Secondary Outcome: Change From Baseline to Month 12 in Cerebral Spinal Fluid for Neurogranin Mean Concentration (pg/mL)
Description: Change from baseline to month 12 in Cerebral Spinal Fluid for Neurogranin Mean Concentration (pg/mL) (samples stored at -70 degrees Celsius; assays performed at Abilene Christian University Bioanalytics Laboratory)
Time Frame: Day 1 to Month 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 18
pg/mL | -115.15 (237.256)

14. Secondary Outcome: Change From Baseline to Month 12 in Cerebral Spinal Fluid for Neurofilament Light Chain Protein Mean Concentration (pg/mL)
Description: Change from baseline to month 12 in Cerebral Spinal Fluid for Neurofilament Light Chain Protein Mean Concentration (pg/mL) (samples stored at -70 degrees Celsius; assays performed at Abilene Christian University Bioanalytics Laboratory)
Time Frame: Day 1 to Month 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 18
pg/mL | -10.00 (95.504)

15. Secondary Outcome: Change From Baseline to Month 12 in Cerebral Spinal Fluid for Glial Fibrillary Acidic Protein Mean Concentration (pg/mL)
Description: Change from baseline to month 12 in Cerebral Spinal Fluid for Glial Fibrillary Acidic Protein Mean Concentration (pg/mL) (samples stored at -70 degrees Celsius; assays performed at Abilene Christian University Bioanalytics Laboratory)
Time Frame: Day 1 to Month 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Simufilam 100 mg Oral Tablets
Number analyzed (Participants) | 18
pg/mL | -84.946 (118.736)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Placebo: Subjects from Month 12 to Month 18 that were taking placebo.
  Placebo: Matching placebo oral tablets administered b.i.d.
- Simufilam: All subjects during day 1 to month 12 (Open-label simufilam), all subjects during month 18 to month 24 (Open-label simufilam), and subjects that were taking simufilam from month 12 to month 18.
  Simufilam 100 mg oral tablet: Simufilam 100 mg oral tablet for b.i.d. administration
Arm/Group | Placebo | Simufilam
All-Cause Mortality (participants affected / at risk) | 1/77 | 1/220
Serious Adverse Events (participants affected / at risk) | 5/77 | 25/220
Other Adverse Events (participants affected / at risk) | 12/77 | 113/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | Simufilam (N=220)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bursitis infective staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=77) | Simufilam (N=220)
COVID-19 (Infections and infestations) | 4 (4) | 26 (26)
Urinary tract infection (Infections and infestations) | 3 (3) | 22 (22)
Headache (Nervous system disorders) | 1 (1) | 19 (19)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 14 (14)
Hypertension (Vascular disorders) | 1 (1) | 13 (13)
Anxiety (Psychiatric disorders) | 1 (1) | 13 (13)
Insomnia (Psychiatric disorders) | 2 (2) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT04388254/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT04388254/SAP_002.pdf